CLINICAL TRIAL: NCT07126626
Title: Multi-center Prospective Validation of the SPOT-MAS Lung Test Using Circulating Tumor DNA for the Detection of Lung Cancer
Brief Title: Validation of the SPOT-MAS Lung Test Using Circulating Tumor DNA for the Detection of Lung Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: Gene Solutions (Industry)
Responsible Party: Sponsor
Other Study IDs: LUNGCARE
Record Dates: First submitted 2025-07-11; First posted 2025-08-17 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Lung Diseases; Lung Cancer Screening
Keywords: SPOT-MAS Lung Test
MeSH Terms: conditions — Lung Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Cohort A 10mL blood sample is collected from eligible participants who have lung cancer screening and are indicated for routine LDCT or NCCT at the enrollment date, for the SPOT-MAS LUNG (SML) test. The blood sample will be transported to the central laboratory of the Institute of Medical Genetics (IMG)
  Cohort B:
  10mL blood sample is collected from eligible participants, who have LDCT or NCCT or CECT results of Lung-RADS 4, valid within 30 days counted from the enrollment date, for the SPOT-MAS LUNG (SML) test. The blood sample will be transported to the central laboratory of the Institute of Medical Genetics (IMG) for plasma separation. The separated plasma will be stored frozen (-80°C) until used for cfDNA extraction and subsequent analytical steps of the SML test procedure.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is an observational clinical trial, aiming to evaluate the efficacy of the SPOTMAS LUNG (SML) test compared to Low dose CTScan (LDCT)/None contrast CTScan (NCCT) in two distinct risk populations:

* Cohort A: To demonstrate that SML is concordant with LDCT/NCCT in general population lung cancer screening, including low-risk (LRs0-1-2), intermediate-risk (LRs3), and high-risk (LRs4) groups.
* Cohort B: To validate the sensitivity and specificity of SML in the high-risk group (LRs4).

DETAILED DESCRIPTION:
This is a prospective, multi-center cohort study to access the performance of SPOT-MAS Lung (SML) in two different scenarios: lung cancer screening (Cohort A) and lung cancer diagnosis (Cohort B).

Sample size and accuracy analyses were performed independently for the study objectives within each cohort. The minimum sample size for Cohort A is approximately 526 samples. Participants will be randomly selected from the screening population for this study without prior LDCT classification criteria. The minimum sample size for Cohort B is approximately 658 samples. Participants will be selected from individuals who have undergone LDCT/NCCT with LUNG-RADS 4 results.

Each Cohort A or B requires a 50% proportion of smokers and 50% of never-smokers or light-smokers, 10mL blood sample and LDCT/NCCT are collected.

Cohort A: According to current lung cancer screening and diagnosis guidelines, volunteers will undergo the following imaging methods:

Lung-RADS 3: Recommended to have a repeat LDCT after 6 and 12 months. Lung-RADS 0-1-2: Recommended to have a repeat LDCT after 12 months. Lung-RADS 4: Recommended to have contrast-enhanced computed tomography (CECT). Cohort B: According to current lung cancer screening and diagnosis guidelines, the Lung-RADS 4 group will be recommended for contrast-enhanced computed tomography (CECT).

Cohort A and B:

If CECT results show a lesion ≥8mm in the lung, biopsy is recommended, and histopathological results evaluated.

* If histopathology is malignant/confirms cancer: proceed with treatment. Treatment costs ARE NOT covered by the study.
* If histopathology is benign: repeat LDCT after 12 months. If CECT results show a lesion <8mm in the lung, or no lesion is seen in the lung, repeat LDCT after 12 months.

LDCT or CECT fee in Month 6 and Month 12 will be covered by this study.

ELIGIBILITY:
Inclusion Criteria:

Cohort A

1. Volunteers (participants) aged 50-80 years at the time of consent.

   1. 50% smokers with a smoking history of 20 pack-years who currently smoke or have quit within the past 15 years.
   2. 50% never-smokers or light smokers (< 20 pack-years or quit > 15 years) who are first- or second-degree relatives of LC patients.
2. Willing to undergo LDCT/NCCT of the chest for lung cancer screening.
3. Willing to consent to an investigational blood draw during the index LDCT/NCCT screening visit and before any invasive procedures or treatment for lung cancer diagnosis.
4. Willing to consent to a 1-year follow-up and additional follow-ups as per protocol.

Cohort B

1. Subjects aged 50-80 years at the time of consent.

   1. 50% smokers with a smoking history of 20 pack-years who currently smoke or have quit within the past 15 years.
   2. 50% never-smokers or light smokers (< 20 pack-years or quit > 15 years) who are first- or second-degree relatives of LC patients.
2. Have undergone LDCT/NCCT of the chest for lung cancer screening/diagnosis, including only high-risk lesions (LUNG-RADS 4).
3. Willing to consent to an investigational blood draw before any invasive procedures (CECT/PET-CT/biopsy) or treatment for lung cancer diagnosis.
4. Willing to consent to a 1-year follow-up and additional follow-ups as per protocol.

Exclusion Criteria for both Cohort A and Cohort B

1. Subject has a health problem that substantially limits life expectancy and/or the ability or willingness to have curative lung surgery.
2. Subject is undergoing CECT for investigation of highly suspicious symptoms for lung cancer.
3. Pre-existing or history of lung cancer.
4. History of any malignancy (subjects who have undergone surgical removal of skin squamous cell cancer may be enrolled provided the procedure was completed at least 12 months prior to the date of provision of informed consent for the study).
5. Currently taking any anti-neoplastic or disease-modifying anti-rheumatic drugs.
6. Currently receiving treatment for pneumonia.
7. Any major physical trauma (e.g., disruption of tissue, surgery, organ transplant, blood product transfusion) within the 30 days leading up to the provision of informed consent.
8. Known medical condition which, in the opinion of the investigator, should preclude enrollment into the study.
9. Participation in a clinical research study in which an experimental medication and/or medical procedure has been administered or may be administered within the 30 days leading up to providing informed consent or may be administered through the time of subject screening.

   -

   Exclusion Criteria:

   -

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cohort A: Patients visit the hospital and are screened according to inclusion/exclusion criteria and are indicated for routine LDCT or NCCT (Enrollment Date D1, results unknown).
  Cohort B: Patients visit the hospital and are screened according to inclusion/exclusion criteria and have LDCT or NCCT or CECT results of Lung-RADS 4, valid within 30 days up to the study enrollment date.
Sampling Method: Probability Sample
Enrollment: 1184 (Estimated)
Dates: Start 2025-08-18 (Estimated); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
The overall objective of this study is to assess the performance of SPOT-MAS LUNG (SML) in two different scenarios: lung cancer screening (Cohort A) and lung cancer diagnosis (Cohort B). | 24 months
  Cohort A • Characteristics: Screening population, including low-risk (LRs0-1-2), intermediate-risk (LRs3), and high-risk (LRs4) patients, taken 10mL blood for SML test.
  Cohort B • Characteristics: High-risk patients (LRs 4), taken 10mL blood for SML test.

SECONDARY OUTCOMES:
Cohort A: To demonstrate that SML is concordant with LDCT/NCCT in the screening population. Cohort B: To assess the specificity and sensitivity of SML in detecting LC in patients with LRs4. | 24 months
  Cohort A: The objective of the study is to demonstrate that SML and LDCT have a high level of agreement, with a Cohen's Kappa coefficient greater than 0.81.
  * Endpoint: The level of agreement between SML and LDCT/NCCT. Cohort B: In a previous case-control study, SML demonstrated a specificity of 92% and a sensitivity of 90% [9]. Thus, this study will be considered successful if the lower-bound of the two-sided 95% Wilson CI of SM for LC sensitivity exceeds 80% and the lower-bound of the two-sided 95% Wilson CI of SM for LC specificity exceeds 82%.
  * Endpoint: Specificity and sensitivity of SML.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Genetics Institute, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Infante MV, Cardillo G. Lung cancer screening in never-smokers: facts and remaining issues. Eur Respir J. 2020 Nov 12;56(5):2002949. doi: 10.1183/13993003.02949-2020. Print 2020 Nov. No abstract available. PMID 33184102
- [Background] Kocher Wulfeck M, Plesner S, Herndon JE 2nd, Christensen JD, Patz EF Jr. Characterizing Lung-RADS category 4 lesions in a university lung cancer screening program. Lung Cancer. 2023 Dec;186:107420. doi: 10.1016/j.lungcan.2023.107420. Epub 2023 Nov 10. PMID 37956610
- [Background] Schulz KF, Grimes DA. Case-control studies: research in reverse. Lancet. 2002 Feb 2;359(9304):431-4. doi: 10.1016/S0140-6736(02)07605-5. PMID 11844534
- [Background] https://doi.org/10.1158/2159-8290.CD-24-0519
- [Background] Hu X, Luo K, Shi H, Yan X, Huang R, Zhao B, Zhang J, Xie D, Zhang W. Integrated 5-hydroxymethylcytosine and fragmentation signatures as enhanced biomarkers in lung cancer. Clin Epigenetics. 2022 Jan 24;14(1):15. doi: 10.1186/s13148-022-01233-7. PMID 35073982
- [Background] Guo W, Chen X, Liu R, Liang N, Ma Q, Bao H, Xu X, Wu X, Yang S, Shao Y, Tan F, Xue Q, Gao S, He J. Sensitive detection of stage I lung adenocarcinoma using plasma cell-free DNA breakpoint motif profiling. EBioMedicine. 2022 Jul;81:104131. doi: 10.1016/j.ebiom.2022.104131. Epub 2022 Jun 30. PMID 35780566
- [Background] http://dx.doi.org/10.1002/mco2.766
- [Background] Jenkins S, Yang JC, Ramalingam SS, Yu K, Patel S, Weston S, Hodge R, Cantarini M, Janne PA, Mitsudomi T, Goss GD. Plasma ctDNA Analysis for Detection of the EGFR T790M Mutation in Patients with Advanced Non-Small Cell Lung Cancer. J Thorac Oncol. 2017 Jul;12(7):1061-1070. doi: 10.1016/j.jtho.2017.04.003. Epub 2017 Apr 17. PMID 28428148
- [Background] Mouliere F, Chandrananda D, Piskorz AM, Moore EK, Morris J, Ahlborn LB, Mair R, Goranova T, Marass F, Heider K, Wan JCM, Supernat A, Hudecova I, Gounaris I, Ros S, Jimenez-Linan M, Garcia-Corbacho J, Patel K, Ostrup O, Murphy S, Eldridge MD, Gale D, Stewart GD, Burge J, Cooper WN, van der Heijden MS, Massie CE, Watts C, Corrie P, Pacey S, Brindle KM, Baird RD, Mau-Sorensen M, Parkinson CA, Smith CG, Brenton JD, Rosenfeld N. Enhanced detection of circulating tumor DNA by fragment size analysis. Sci Transl Med. 2018 Nov 7;10(466):eaat4921. doi: 10.1126/scitranslmed.aat4921. PMID 30404863
- [Background] Snyder MW, Kircher M, Hill AJ, Daza RM, Shendure J. Cell-free DNA Comprises an In Vivo Nucleosome Footprint that Informs Its Tissues-Of-Origin. Cell. 2016 Jan 14;164(1-2):57-68. doi: 10.1016/j.cell.2015.11.050. PMID 26771485
- [Background] Weiss G, Schlegel A, Kottwitz D, Konig T, Tetzner R. Validation of the SHOX2/PTGER4 DNA Methylation Marker Panel for Plasma-Based Discrimination between Patients with Malignant and Nonmalignant Lung Disease. J Thorac Oncol. 2017 Jan;12(1):77-84. doi: 10.1016/j.jtho.2016.08.123. Epub 2016 Aug 18. PMID 27544059
- [Background] Johnson DA, Barclay RL, Mergener K, Weiss G, Konig T, Beck J, Potter NT. Plasma Septin9 versus fecal immunochemical testing for colorectal cancer screening: a prospective multicenter study. PLoS One. 2014 Jun 5;9(6):e98238. doi: 10.1371/journal.pone.0098238. eCollection 2014. PMID 24901436
- [Background] Ehrlich M. DNA hypomethylation in cancer cells. Epigenomics. 2009 Dec;1(2):239-59. doi: 10.2217/epi.09.33. PMID 20495664
- [Background] McCabe MT, Brandes JC, Vertino PM. Cancer DNA methylation: molecular mechanisms and clinical implications. Clin Cancer Res. 2009 Jun 15;15(12):3927-37. doi: 10.1158/1078-0432.CCR-08-2784. Epub 2009 Jun 9. PMID 19509173
- [Background] Pecuchet N, Zonta E, Didelot A, Combe P, Thibault C, Gibault L, Lours C, Rozenholc Y, Taly V, Laurent-Puig P, Blons H, Fabre E. Base-Position Error Rate Analysis of Next-Generation Sequencing Applied to Circulating Tumor DNA in Non-Small Cell Lung Cancer: A Prospective Study. PLoS Med. 2016 Dec 27;13(12):e1002199. doi: 10.1371/journal.pmed.1002199. eCollection 2016 Dec. PMID 28027313
- [Background] Filipska M, Rosell R. Mutated circulating tumor DNA as a liquid biopsy in lung cancer detection and treatment. Mol Oncol. 2021 Jun;15(6):1667-1682. doi: 10.1002/1878-0261.12983. Epub 2021 May 26. PMID 33969622
- [Background] Zhao X, Dai F, Mei L, Huang D, Shen X, Zhang H, She X, Ma Z. The Potential Use of Dynamics Changes of ctDNA and cfDNA in the Perioperative Period to Predict the Recurrence Risk in Early NSCLC. Front Oncol. 2021 Jul 16;11:671963. doi: 10.3389/fonc.2021.671963. eCollection 2021. PMID 34336662
- [Background] Zhang X, Li J, Lan X, Li J. Cell-free DNA-associated multi-feature applications in cancer diagnosis and treatment. Vol. 4, Clinical and Translational Discovery. 2024.
- [Background] Volckmar AL, Sultmann H, Riediger A, Fioretos T, Schirmacher P, Endris V, Stenzinger A, Dietz S. A field guide for cancer diagnostics using cell-free DNA: From principles to practice and clinical applications. Genes Chromosomes Cancer. 2018 Mar;57(3):123-139. doi: 10.1002/gcc.22517. Epub 2017 Dec 20. PMID 29205637
- [Background] Qi T, Pan M, Shi H, Wang L, Bai Y, Ge Q. Cell-Free DNA Fragmentomics: The Novel Promising Biomarker. Int J Mol Sci. 2023 Jan 12;24(2):1503. doi: 10.3390/ijms24021503. PMID 36675018
- [Background] Stoecklein NH, Fischer JC, Niederacher D, Terstappen LW. Challenges for CTC-based liquid biopsies: low CTC frequency and diagnostic leukapheresis as a potential solution. Expert Rev Mol Diagn. 2016;16(2):147-64. doi: 10.1586/14737159.2016.1123095. Epub 2015 Dec 16. PMID 26587751
- [Background] Wan S, Kim TH, Smith KJ, Delaney R, Park GS, Guo H, Lin E, Plegue T, Kuo N, Steffes J, Leu C, Simeone DM, Razimulava N, Parikh ND, Nagrath S, Welling TH. New Labyrinth Microfluidic Device Detects Circulating Tumor Cells Expressing Cancer Stem Cell Marker and Circulating Tumor Microemboli in Hepatocellular Carcinoma. Sci Rep. 2019 Dec 9;9(1):18575. doi: 10.1038/s41598-019-54960-y. PMID 31819089
- [Background] Fachin F, Spuhler P, Martel-Foley JM, Edd JF, Barber TA, Walsh J, Karabacak M, Pai V, Yu M, Smith K, Hwang H, Yang J, Shah S, Yarmush R, Sequist LV, Stott SL, Maheswaran S, Haber DA, Kapur R, Toner M. Monolithic Chip for High-throughput Blood Cell Depletion to Sort Rare Circulating Tumor Cells. Sci Rep. 2017 Sep 7;7(1):10936. doi: 10.1038/s41598-017-11119-x. PMID 28883519
- [Background] Alix-Panabieres C, Pantel K. Clinical Applications of Circulating Tumor Cells and Circulating Tumor DNA as Liquid Biopsy. Cancer Discov. 2016 May;6(5):479-91. doi: 10.1158/2159-8290.CD-15-1483. Epub 2016 Mar 11. PMID 26969689
- [Background] Schrag D, Beer TM, McDonnell CH 3rd, Nadauld L, Dilaveri CA, Reid R, Marinac CR, Chung KC, Lopatin M, Fung ET, Klein EA. Blood-based tests for multicancer early detection (PATHFINDER): a prospective cohort study. Lancet. 2023 Oct 7;402(10409):1251-1260. doi: 10.1016/S0140-6736(23)01700-2. PMID 37805216
- [Background] Vacante M, Ciuni R, Basile F, Biondi A. The Liquid Biopsy in the Management of Colorectal Cancer: An Overview. Biomedicines. 2020 Aug 26;8(9):308. doi: 10.3390/biomedicines8090308. PMID 32858879
- [Background] Hirahata T, Ul Quraish R, Quraish AU, Ul Quraish S, Naz M, Razzaq MA. Liquid Biopsy: A Distinctive Approach to the Diagnosis and Prognosis of Cancer. Cancer Inform. 2022 Feb 7;21:11769351221076062. doi: 10.1177/11769351221076062. eCollection 2022. PMID 35153470
- [Background] Duy TH, Thọ NV, Linh LTM, Hoàng PM, Tố TT, Thùy BTC, Ngọc NTM, Phương NM. Tỷ lệ và đặc điểm ung thư phổi ở nhóm đối tượng nguy cơ cao đánh giá thông qua chụp cắt lớp vi tính lồng ngực liều thấp. Tạp chí Y học Việt Nam. 2024;537(1).
- [Background] Hà HTN, Tiến ĐD, Khoan LT. Nghiên cứu giá trị của cắt lớp vi tính ngực liều thấp trong phát hiện sớm các nốt mở phổi ác . Tạp Chí Y Dược Huế. 2020;10(4):7-15.
- [Background] Đặng ĐP, Ngô QB, Đinh HV, Nguyễn QĐ. Giá trị của phân loại lung-rads trong chẩn đoán ung thư phổi với nốt mờ đơn độc. Tạp chí Y học Việt Nam. 2022;520(1A).
- [Background] Torres S, Gonzalez A, Cunquero Tomas AJ, Calabuig Farinas S, Ferrero M, Mirda D, Sirera R, Jantus-Lewintre E, Camps C. A profile on cobas(R) EGFR Mutation Test v2 as companion diagnostic for first-line treatment of patients with non-small cell lung cancer. Expert Rev Mol Diagn. 2020 Jun;20(6):575-582. doi: 10.1080/14737159.2020.1724094. Epub 2020 Feb 20. PMID 32011193
- [Background] Winokur RS, Pua BB, Sullivan BW, Madoff DC. Percutaneous lung biopsy: technique, efficacy, and complications. Semin Intervent Radiol. 2013 Jun;30(2):121-7. doi: 10.1055/s-0033-1342952. PMID 24436527
- [Background] Yasufuku K, Pierre A, Darling G, de Perrot M, Waddell T, Johnston M, da Cunha Santos G, Geddie W, Boerner S, Le LW, Keshavjee S. A prospective controlled trial of endobronchial ultrasound-guided transbronchial needle aspiration compared with mediastinoscopy for mediastinal lymph node staging of lung cancer. J Thorac Cardiovasc Surg. 2011 Dec;142(6):1393-400.e1. doi: 10.1016/j.jtcvs.2011.08.037. Epub 2011 Oct 2. PMID 21963329
- [Background] Wimaleswaran H, Farmer MW, Irving LB, Jennings BR, Steinfort DP. Pulmonologist-performed transoesophageal sampling for lung cancer staging using an endobronchial ultrasound video-bronchoscope: an Australian experience. Intern Med J. 2017 Feb;47(2):205-210. doi: 10.1111/imj.13330. PMID 27860078
- [Background] Cham MD, Henschke CI, Yankelevitz DF. The radiologist's role in pathologic diagnosis of small lung nodules: radiographic methods of tissue acquisition. Current Challenges in Thoracic Surgery. 2022;4.
- [Background] Silvestri GA, Goldman L, Tanner NT, Burleson J, Gould M, Kazerooni EA, Mazzone PJ, Rivera MP, Doria-Rose VP, Rosenthal LS, Simanowith M, Smith RA, Fedewa S. Outcomes From More Than 1 Million People Screened for Lung Cancer With Low-Dose CT Imaging. Chest. 2023 Jul;164(1):241-251. doi: 10.1016/j.chest.2023.02.003. Epub 2023 Feb 10. PMID 36773935
- [Background] Meza R, Jeon J, Toumazis I, Ten Haaf K, Cao P, Bastani M, Han SS, Blom EF, Jonas DE, Feuer EJ, Plevritis SK, de Koning HJ, Kong CY. Evaluation of the Benefits and Harms of Lung Cancer Screening With Low-Dose Computed Tomography: Modeling Study for the US Preventive Services Task Force. JAMA. 2021 Mar 9;325(10):988-997. doi: 10.1001/jama.2021.1077. PMID 33687469
- [Background] Reinke LF, Feemster LC, Backhus LM, Gylys-Colwell I, Au DH. Assessment and Management of Symptoms for Outpatients Newly Diagnosed With Lung Cancer. Am J Hosp Palliat Care. 2016 Mar;33(2):178-83. doi: 10.1177/1049909114557635. Epub 2014 Nov 5. PMID 25376224
- [Background] Butler SJ, Louie AV, Sutradhar R, Paszat L, Brooks D, Gershon AS. Impact of chronic obstructive pulmonary disease on lung cancer symptom burden: a population-based study in Ontario, Canada. Transl Lung Cancer Res. 2023 Nov 30;12(11):2260-2274. doi: 10.21037/tlcr-23-560. Epub 2023 Nov 28. PMID 38090519
- [Background] Wakelee HA, Chang ET, Gomez SL, Keegan TH, Feskanich D, Clarke CA, Holmberg L, Yong LC, Kolonel LN, Gould MK, West DW. Lung cancer incidence in never smokers. J Clin Oncol. 2007 Feb 10;25(5):472-8. doi: 10.1200/JCO.2006.07.2983. PMID 17290054
- [Background] Sun S, Schiller JH, Gazdar AF. Lung cancer in never smokers--a different disease. Nat Rev Cancer. 2007 Oct;7(10):778-90. doi: 10.1038/nrc2190. PMID 17882278
- [Background] Pelosof L, Ahn C, Gao A, Horn L, Madrigales A, Cox J, McGavic D, Minna JD, Gazdar AF, Schiller J. Proportion of Never-Smoker Non-Small Cell Lung Cancer Patients at Three Diverse Institutions. J Natl Cancer Inst. 2017 Jan 28;109(7):djw295. doi: 10.1093/jnci/djw295. Print 2017 Jan. PMID 28132018
- [Background] Zeng Q, Vogtmann E, Jia MM, Parascandola M, Li JB, Wu YL, Feng QF, Zou XN. Tobacco smoking and trends in histological subtypes of female lung cancer at the Cancer Hospital of the Chinese Academy of Medical Sciences over 13 years. Thorac Cancer. 2019 Aug;10(8):1717-1724. doi: 10.1111/1759-7714.13141. Epub 2019 Jul 10. PMID 31293059
- [Background] Doğan C. Different Characteristics in Lung Cancer Patients Between Age Groups Under 55 and Over 55 Years of Age? South Clin Istanb Eurasia. 2017;
- [Background] Tarigan SP, Soeroso NN, Tumanggor CAK, Gani S, Pradana A. Clinical Profile of Male Patients with Non-Small Cell Lung Cancer in Adam Malik General Hospital, Medan, Indonesia. Open Access Maced J Med Sci. 2019 Aug 29;7(16):2612-2614. doi: 10.3889/oamjms.2019.404. eCollection 2019 Aug 30. PMID 31777616
- [Background] Barta JA, Zinner RG, Unger M. Lung Cancer in the Older Patient. Clin Geriatr Med. 2017 Nov;33(4):563-577. doi: 10.1016/j.cger.2017.06.008. Epub 2017 Aug 19. PMID 28991651
- [Background] Torre LA, Siegel RL, Jemal A. Lung Cancer Statistics. Adv Exp Med Biol. 2016;893:1-19. doi: 10.1007/978-3-319-24223-1_1. PMID 26667336
- [Background] Krewski D, Lubin JH, Zielinski JM, Alavanja M, Catalan VS, Field RW, Klotz JB, Letourneau EG, Lynch CF, Lyon JI, Sandler DP, Schoenberg JB, Steck DJ, Stolwijk JA, Weinberg C, Wilcox HB. Residential radon and risk of lung cancer: a combined analysis of 7 North American case-control studies. Epidemiology. 2005 Mar;16(2):137-45. doi: 10.1097/01.ede.0000152522.80261.e3. PMID 15703527
- [Background] van Loon AJ, Kant IJ, Swaen GM, Goldbohm RA, Kremer AM, van den Brandt PA. Occupational exposure to carcinogens and risk of lung cancer: results from The Netherlands cohort study. Occup Environ Med. 1997 Nov;54(11):817-24. doi: 10.1136/oem.54.11.817. PMID 9538355
- [Background] Pope CA 3rd, Burnett RT, Thun MJ, Calle EE, Krewski D, Ito K, Thurston GD. Lung cancer, cardiopulmonary mortality, and long-term exposure to fine particulate air pollution. JAMA. 2002 Mar 6;287(9):1132-41. doi: 10.1001/jama.287.9.1132. PMID 11879110
- [Background] Taylor R, Najafi F, Dobson A. Meta-analysis of studies of passive smoking and lung cancer: effects of study type and continent. Int J Epidemiol. 2007 Oct;36(5):1048-59. doi: 10.1093/ije/dym158. Epub 2007 Aug 9. PMID 17690135
- [Background] Expert Panel on Thoracic Imaging:; de Groot PM, Chung JH, Ackman JB, Berry MF, Carter BW, Colletti PM, Hobbs SB, McComb BL, Movsas B, Tong BC, Walker CM, Yom SS, Kanne JP. ACR Appropriateness Criteria(R) Noninvasive Clinical Staging of Primary Lung Cancer. J Am Coll Radiol. 2019 May;16(5S):S184-S195. doi: 10.1016/j.jacr.2019.02.008. PMID 31054745
- [Background] US Preventive Services Task Force; Krist AH, Davidson KW, Mangione CM, Barry MJ, Cabana M, Caughey AB, Davis EM, Donahue KE, Doubeni CA, Kubik M, Landefeld CS, Li L, Ogedegbe G, Owens DK, Pbert L, Silverstein M, Stevermer J, Tseng CW, Wong JB. Screening for Lung Cancer: US Preventive Services Task Force Recommendation Statement. JAMA. 2021 Mar 9;325(10):962-970. doi: 10.1001/jama.2021.1117. PMID 33687470
- [Background] Freedman ND, Abnet CC, Caporaso NE, Fraumeni JF Jr, Murphy G, Hartge P, Hollenbeck AR, Park Y, Shiels MS, Silverman DT. Impact of changing US cigarette smoking patterns on incident cancer: risks of 20 smoking-related cancers among the women and men of the NIH-AARP cohort. Int J Epidemiol. 2016 Jun;45(3):846-56. doi: 10.1093/ije/dyv175. Epub 2015 Sep 27. PMID 26411408
- [Background] Herbst RS, Morgensztern D, Boshoff C. The biology and management of non-small cell lung cancer. Nature. 2018 Jan 24;553(7689):446-454. doi: 10.1038/nature25183. PMID 29364287
- [Background] Bray F, Laversanne M, Sung H, Ferlay J, Siegel RL, Soerjomataram I, Jemal A. Global cancer statistics 2022: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2024 May-Jun;74(3):229-263. doi: 10.3322/caac.21834. Epub 2024 Apr 4. PMID 38572751
- [Background] Nguyen VTC, Nguyen TH, Doan NNT, Pham TMQ, Nguyen GTH, Nguyen TD, Tran TTT, Vo DL, Phan TH, Jasmine TX, Nguyen VC, Nguyen HT, Nguyen TV, Nguyen THH, Huynh LAK, Tran TH, Dang QT, Doan TN, Tran AM, Nguyen VH, Nguyen VTA, Ho LMQ, Tran QD, Pham TTT, Ho TD, Nguyen BT, Nguyen TNV, Nguyen TD, Phu DTB, Phan BHH, Vo TL, Nai THT, Tran TT, Truong MH, Tran NC, Le TK, Tran THT, Duong ML, Bach HPT, Kim VV, Pham TA, Tran DH, Le TNA, Pham TVN, Le MT, Vo DH, Tran TMT, Nguyen MN, Van TTV, Nguyen AN, Tran TT, Tran VU, Le MP, Do TT, Phan TV, Nguyen HL, Nguyen DS, Cao VT, Do TT, Truong DK, Tang HS, Giang H, Nguyen HN, Phan MD, Tran LS. Multimodal analysis of methylomics and fragmentomics in plasma cell-free DNA for multi-cancer early detection and localization. Elife. 2023 Oct 11;12:RP89083. doi: 10.7554/eLife.89083. PMID 37819044
- [Background] Wang S, Meng F, Li M, Bao H, Chen X, Zhu M, Liu R, Xu X, Yang S, Wu X, Shao Y, Xu L, Yin R. Multidimensional Cell-Free DNA Fragmentomic Assay for Detection of Early-Stage Lung Cancer. Am J Respir Crit Care Med. 2023 May 1;207(9):1203-1213. doi: 10.1164/rccm.202109-2019OC. PMID 36346614
- [Background] http://dx.doi.org/10.1056/NEJMoa1102873
- [Background] Sagawa M, Sakurada A, Ashizawa K, Maeda S, Nakayama T, Oikado K, Gemba K, Kobayashi T, Torii Y, Takenaka D, Maruyama Y, Mitomo H, Murota M, Yanagawa M, Shibuya K, Sobue T, Harada M, Miura H. Revision of the Lung Cancer Screening Guidelines in 2022. Japanese Journal of Lung Cancer. 2022;62(5).
- [Background] Chinese Expert Group on Early Diagnosis and Treatment of Lung Cancer; China Lung Oncology Group. [China National Lung Cancer Screening Guideline with Low-dose Computed Tomography (2023 Version)]. Zhongguo Fei Ai Za Zhi. 2023 Jan 20;26(1):1-9. doi: 10.3779/j.issn.1009-3419.2023.102.10. Chinese. PMID 36792074
- [Background] Chapter of Respiratory Physicians C of PA of MS. Lung Cancer Screening in Singapore: Professional Guidelines. Singapore; 2025 Jan
- [Background] Lam DC, Liam CK, Andarini S, Park S, Tan DSW, Singh N, Jang SH, Vardhanabhuti V, Ramos AB, Nakayama T, Nhung NV, Ashizawa K, Chang YC, Tscheikuna J, Van CC, Chan WY, Lai YH, Yang PC. Lung Cancer Screening in Asia: An Expert Consensus Report. J Thorac Oncol. 2023 Oct;18(10):1303-1322. doi: 10.1016/j.jtho.2023.06.014. Epub 2023 Jun 28. PMID 37390982